CLINICAL TRIAL: NCT02174757
Title: A Comparative Evaluation of the Effect of Probiotic Inersan and Doxycycline on Chronic Periodontitis - A Clinical and Microbiological Study
Brief Title: Effect of Probiotic Inersan and Doxycycline in Chronic Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CD Pharma India Pvt. Ltd. (Industry)
Collaborators: Sree Mookambika Institute of Dental Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUL_SMIDS_PERIO_01
Record Dates: First submitted 2014-06-19; First posted 2014-06-26 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inersan (Experimental): Inersan - 2 Lozenges daily (one lozenge in morning and one lozenge in night) for 2 weeks. Each lozenge contains at least 1 billion CFU of Lactobacillus brevis CD2.
  Interventions: Drug: Inersan
- Inersan and Doxycycline together (Experimental): Doxycycline: 1 Tablet once daily (in afternoon) for 2 weeks. Each tablet contains 100 mg Doxycycline.
  Inersan - 2 Lozenges daily (one lozenge in morning and one lozenge in night) for 2 weeks. Each lozenge contains at least 1 billion CFU of Lactobacillus brevis CD2.
  Interventions: Drug: Inersan; Drug: Doxycycline
- Doxycycline (Active Comparator): Doxycycline: 1 Tablet once daily (in afternoon) for 2 weeks. Each tablet contains 100 mg Doxycycline.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Inersan — Probiotic
  Other Names: Each lozenge contains not less than 1 billion CFU of Lactobacillus brevis CD2
  Arms: Inersan; Inersan and Doxycycline together
Drug: Doxycycline — Antibiotic
  Other Names: Each tablet contains 100 mg of Doxycycline
  Arms: Doxycycline; Inersan and Doxycycline together

SUMMARY:
Periodontitis is a multifactorial disease that can lead to the destruction of supporting tissues of the teeth resulting in pocket formation, recession or both. Since the primary etiological factors for periodontal disease are bacteria in supra and sub gingival biofilm, efforts for disease prevention and treatment are mainly focused on pathogen reduction and strengthening of epithelial barrier, thus contributing to decreased susceptibility to infection. Due to emergence of antibiotic resistance and frequent recolonization of treated sites with pathogenic bacteria, there was need for a new treatment paradigm to be introduced to periodontal disease. The need was fulfilled by the introduction of Probiotics and Bacterial Replacement Therapy. The term probiotic is derived from the Greek, meaning "for life" are microorganisms proven to exert health promoting influences in humans and animals. Food and Agriculture Organization and WHO have stated that there is potential for probiotic foods to provide health benefits and that specific strains are safe for human use.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects in both sexes
2. Age 25 - 60 yrs
3. Subjects with mild to moderate chronic periodontitis, as defined by probing pocket depths ≥ 5mm in > 30 % of the probing sites
4. Subjects in good general health

Exclusion Criteria:

1. Antibiotic therapy in the past 2 months
2. Allergic to doxycycline or probiotics
3. Subjects with diabetic mellitus, hypertension and psychiatric disorders
4. Subjects who are pregnant/ lactating
5. Smokers and/or alcoholics
6. Subjects who have undergone any periodontal therapy within last 6 months.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Improvement in periodontal clinical indices | 4 weeks
  Improvement in periodontal clinical indices, namely, Gingival Index (GI), Probing Pocket Depth (PPD), Plaque Index (PI) and Clinical Attachment level (CAL)

SECONDARY OUTCOMES:
Improvement in microbiological indices | 4 weeks
  Changes in salivary count of Lactobacilli and Porphyromonas gingivalis

CONTACTS AND LOCATIONS:
Overall Officials: Arya K.S., BDS, Principal Investigator — Sree Mookambika Institute of Dental Sciences; Elizabeth Koshi, MDS, Study Director — Sree Mookambika Institute of Dental Sciences; Arun Sadasivan, MDS, Principal Investigator — Sree Mookambika Institute of Dental Sciences
Locations (1):
- Dept. of Periodontics and Implantology, Sree Mookambika Institute of Dental Sciences, Kulasegaram, Tamil Naidu, India